CLINICAL TRIAL: NCT05611476
Title: Cognitive Muscular Therapy for Low Back Pain
Acronym: CMT-LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Responsible Party: Principal Investigator, Stephen Preece, Professor of Biomechanics and Rehabilitation, University of Salford
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMT-LBP-6581
Record Dates: First submitted 2022-11-01; First posted 2022-11-10 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Low Back Pain; Chronic Pain; Muscle Tightness
Keywords: Psychologically informed physiotherapy; Electromyography biofeedback; Cognitive Muscular Therapy
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: The primary aim is to develop the intervention. We will do this through delivery of the intervention to three waves of patients. After each of the first two waves, the intervention will be adapted based on participant feedback
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): This group will receive Cognitive Muscular Therapy for low back pain
  Interventions: Behavioral: Cognitive Muscular Therapy for low back pain

INTERVENTIONS:
Behavioral: Cognitive Muscular Therapy for low back pain — Psychologically informed physiotherapy which used biofeedback training to reduce muscle overactivity and improve postural control

SUMMARY:
The primary aim of this study is to adapt Cognitive Muscular Therapy so that it can be used to manage chronic low back pain. A secondary aim is to understand the potential therapeutic benefit of this intervention.

DETAILED DESCRIPTION:
There is evidence that people with chronic low back pain (LBP) demonstrate muscle overactivity during functional tasks when compared to healthy controls. Interestingly, this increased activity of the low back and trun, muscles has been associated with increased sensitivity to pain. It has also been shown that people with chronic LBP exhibit alterations in functional movement patterns and postures when compared to healthy people. Such alterations may be a direct result of increased stiffness in the spine which results from muscle overactivity. Psychosocial physiotherapy techniques for LBP are gaining widescale acceptance. However, these approaches are often combined with strengthening exercises, and not specifically aimed at reducing muscle overactivity. Therefore, there is a need for research into interventions for chronic LBP which integrate psychologically informed practice with training to reduce muscle overactivity.

The investigators have developed a new treatment for people with knee osteoarthritis, known as Cognitive Muscular Therapy (CMT). CMT is a form of psychologically informed physiotherapy which uses biofeedback training to reduce muscle overactivity and therefore lower the mechanical stress on the knee. CMT is delivered through five sequential intervention components and teaches patients to think and respond differently to pain, to improve postural control and to perform functional movements, such as walking, with less muscle tension. See the dedicated website for further details (https://hub.salford.ac.uk/cognitive-muscular-therapy/). Given the strong focus on postural control, the investigators are confident that CMT can be adapted and used to treat other chronic musculoskeletal conditions, such as LBP. In this project, the investigators will map changes to the five CMT intervention components. The intervention will then be delivered to patients with chronic low back pain, after which the investigators will seek to understand participant perceptions of the new treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Above 18 years old
2. Speak and understand English sufficient to read the information sheet and sign the consent form
3. Ability to walk without an assistive device for at least 100m (to ensure patients have sufficient mobility to be able to complete the intervention)
4. Low back pain for at least three months' duration
5. Currently scoring 4 or more on the Roland disability scale

Exclusion Criteria:

1. Dementia or other major cognitive impairment
2. Red flags (specific causes of LBP, such as acute disc prolapse with radicular pain, or other serious pathology)
3. Pregnancy
4. History of serious spinal injury (fractures, spinal cord injury)
5. BMI >33 (as EMG measurement is not possible in people with higher BMI)
6. Acute low back pain (Onset less than 3 months)
7. Any systemic inflammatory disorders, such as rheumatoid arthritis
8. Any balance disorders which may increase the risk of a fall

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Change in Rowland Morris Disability questionnaire | Change from baseline to 2 months
  Used to capture pain/disability associated with low back pain. Score 0-24 (0=no pain, 24=maximum pain)

SECONDARY OUTCOMES:
Change in Pain catastrophizing scale | Change from baseline to 2 months
  Used to capture pain catastrophizing behaviours. Score 0-52 (0=no pain catastrophizing, 52=maximum pain catastrophizing)
Change in Tampa scale of kinesiophobia | Change from baseline to 2 months
  Used to capture kinesiophobia behaviours. Score 17-68 (0=no kinesiophobia, 52=maximum kinesiophobia)
Change in Oswestry disability scale | Change from baseline to 2 months
  Used to capture intensity of low back pain. Score 0-100 (0=no pain)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Salford, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
We may make the clinical data available through a document which will be linked to the journal paper we publish

REFERENCES:
- [Derived] Preece SJ, Smith J, Brookes N, Gates S, Ghio D. Cognitive Muscular Therapy for low back pain: a pilot study. Musculoskelet Sci Pract. 2025 Nov;80:103415. doi: 10.1016/j.msksp.2025.103415. Epub 2025 Sep 13. PMID 40972445
- See also: Description of CMT for knee pain. This will be adapted for low back pain. — https://hub.salford.ac.uk/cognitive-muscular-therapy/